CLINICAL TRIAL: NCT02121821
Title: Impact Evaluation of the Pilot SMS Mother Reminder System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: African Strategies for Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSH-001
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Effects of the SMS Mother Reminder System on Use of Health Care.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): A control group of pregnant women receiving no intervention (i.e. no SMS reminders).
- SMS reminder messages (Experimental): The intervention group will be composed of pregnant women receiving SMS reminder messages via the SMS Mother Reminder system.
  Interventions: Behavioral: SMS reminder messages

INTERVENTIONS:
Behavioral: SMS reminder messages — The study is prospective and interventional comparing differences between pregnant women who receive reminder messages via the SMS Mother Reminder system to those who are not. Pregnant women will be followed from their first ANC visit at a health facility through delivery. The study will examine the effect of the mobile phone intervention on attendance to ANC appointments and IPTP2 coverage. The intervention group will be composed of pregnant women receiving SMS reminder messages in comparison with a control group of pregnant women receiving no intervention (i.e. no SMS reminders).
  Arms: SMS reminder messages

SUMMARY:
The study aims to assess the effects of the SMS Mother Reminder system on use of health care in Uganda. A secondary aim of the study is to determine the behavioral factors and cost-effectiveness, as well as test the usability of the SMS Mother Reminder in Uganda.

DETAILED DESCRIPTION:
USAID/Uganda is commissioning a prospective impact evaluation of the initial SMS component of Uganda's National Health Record Program (NHRP) in order to inform strategic targeting of eHealth and future investments after the pilot phase of the NHRP mobile platform "SMS Mother Reminder". This impact evaluation will be designed to answer the following questions:

Primary evaluation question:

• What is the effect on maternal health outcomes (ANC4 and IPTP2) of the village health teams' use of the SMS Mother Reminder system?

Secondary evaluation questions:

* What factors most influence changes in health workers, village health teams and expectant women's knowledge, attitudes and practices in maternal health?
* To what extent is using the SMS Mother Reminder application to track and inform pregnant women a cost-effective intervention from the perspectives of USAID?
* To what extent can users easily carry out specific tasks (e.g. entering the information of pregnant women) of the SMS Mother Reminder application on mobile devices?

This study is funded by USAID through the African Strategies for Health project.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11454 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
ANC visits | 1 year
  Pregnant women attend 4 Antenatal care visits (ANC)
SP doses | 1 year
  Pregnant women receive at least 2 doses of intermittent preventive treatment of malaria in pregnancy using sulfadoxine-pyrimethamine (SP).

CONTACTS AND LOCATIONS:
Overall Officials: Donald Shepard, Ph.D., Principal Investigator — Brandeis University
Locations (1):
- Gulu District Health Centers, Gulu, Gulu, Uganda